CLINICAL TRIAL: NCT00001243
Title: Effects of Infection With the Human Immunodeficiency Virus on the Development and Function of Bone Marrow Cells
Brief Title: Effects of HIV on the Development and Function of Bone Marrow Cells
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 890035; 89-I-0035
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-12

CONDITIONS: HIV Infection
Keywords: AIDS; Myeloid Progenitors; Monocytes; Plasmid Libraries; Cytokines
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

SUMMARY:
This study will examine the effects of HIV on bone marrow cells. Various types of cells from bone marrow will be studied to learn which cells become infected with HIV, what changes occur in the number of or growth patterns of the cells, what kinds of proteins the cells make in the presence or absence of HIV and whether the cells can function normally.

HIV-infected and non-infected individuals 18 years of age and older may participate in this study.

Participants will undergo the following procedures:

* Blood draw: Blood will be drawn through a needle from a hand or arm vein. About 150 milliliters (10 tablespoons) will be collected each time. No more than 450 ml (30 tablespoons) will be taken over a 6-week period.
* Bone marrow aspirate: Bone marrow will be drawn from the hipbone. For this procedure, a local anesthetic is injected in the skin over the hipbone. A small needle is put about 1/2-inch through the shell of the bone and about 3 to 4 teaspoons of marrow are drawn from the cavity into a syringe.

White cells from marrow of uninfected individuals may be infected with HIV in the laboratory and grown over time for study. Alternatively, uninfected cells may be used as controls to compare with cells from HIV-infected individuals.

White cells from marrow of HIV-infected individuals will be grown in the laboratory and studied in comparison with cells from uninfected individuals. Or, bone marrow cells may be injected into immune-deficient mice to try to develop an animal model for HIV infection. White blood cells will also be studied in the laboratory to learn how the immune system responds to HIV infection.

DETAILED DESCRIPTION:
Hematologic abnormalities occur with high frequency (up to 70% of patients) in human immunodeficiency virus (HIV) infected individuals. The pathogenesis of these abnormalities is not currently understood, although both an abnormal bone marrow environment (e.g., altered growth factor production) and direct infection and dysfunction of progenitor cells themselves have been postulated. Under the current protocol we have studied bone marrow precursor cells from both HIV infected and uninfected individuals and have shown not only that these cells are infectable in vitro with HIV but also infected in vivo in a subpopulation of seropositive individuals. While the effects of HIV infection of precursor cells on subsequent hematopoietic potential is not completely understood, we could not show a clear correlation between in vivo infection of these cells and suppressed hematopoiesis. It seems clear from this study and others that other alterations within the bone marrow environment must play a role in the clinically observed hematologic abnormalities. We therefore wish to continue our studies to elucidate the relative contributions of direct infection of myeloid progenitor cells and alterations in bone marrow environment in the pathology seen in HIV infected individuals. Understanding the pathogenesis of abnormal hematopoiesis in HIV infection will allow investigators to design appropriate therapeutic strategies. Using recently developed techniques we also wish to use bone marrow cells from HIV infected individuals to establish antibody libraries. This will allow the study of immunologically important epitopes on the HIV virion with potential impact on the subsequent design of HIV vaccines or introduction of passive immunotherapy. Thirdly, research in the field of HIV has been hampered by the lack of an appropriate animal model. One promising approach is the use of human bone marrow to reconstitute lethally irradiated Balb/c mice. Once the human hematopoietic system is established in the mouse, it may be possible to infect these animals with HIV and study in an in vivo model the effects of infection on hematopoiesis.

ELIGIBILITY:
INCLUSION CRITERIA:

Both HIV seropositive and seronegative individuals.

Have adequate blood counts (HIV positive volunteers: hemoglobin greater than or equal to 9.0 g/dL, HCT greater than or equal to 28%, platelets greater than or equal to 50,000; HIV negative healthy normal volunteers: hemoglobin greater than or equal to 12.5 g/dL, HCT greater than or equal to 38%, platelets greater than or equal to 150,000.

Aged 18 years or older, male or female.

Ability to give informed, written consent.

This protocol was amended in 1990 to allow inclusion of Zairian patients who were studied by the principal investigator on site in Zaire. These marrow aspirations were all performed in March-April 1990 before the current requirements for Multi-site Collaborations were instituted. At this time, no further off-site collaboration will be undertaken under this protocol.

EXCLUSION CRITERIA:

Women who are pregnant.

Patients/volunteers with blood clotting disorders as demonstrated by an elevated PT, PTT or low platelet count (Seropositive: platelets greater than or equal to 50,000; Seronegative: platelets greater than or equal to150,000.

Patients/Volunteers who are taking NSAIDS or other anti-coagulant medication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1989-02; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Folks TM, Kessler SW, Orenstein JM, Justement JS, Jaffe ES, Fauci AS. Infection and replication of HIV-1 in purified progenitor cells of normal human bone marrow. Science. 1988 Nov 11;242(4880):919-22. doi: 10.1126/science.2460922.
- [Background] Donahue RE, Johnson MM, Zon LI, Clark SC, Groopman JE. Suppression of in vitro haematopoiesis following human immunodeficiency virus infection. Nature. 1987 Mar 12-18;326(6109):200-3. doi: 10.1038/326200a0. PMID 2434864
- [Background] Steinberg HN, Crumpacker CS, Chatis PA. In vitro suppression of normal human bone marrow progenitor cells by human immunodeficiency virus. J Virol. 1991 Apr;65(4):1765-9. doi: 10.1128/JVI.65.4.1765-1769.1991. PMID 2002542